CLINICAL TRIAL: NCT02181010
Title: B'More Healthy: Communities for Kids (BHCK)
Brief Title: B'More Healthy; Communities for Kids (BHCK)
Acronym: BHCK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 111189
Record Dates: First submitted 2014-06-20; First posted 2014-07-03 (Estimated); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Obesity
Keywords: African American; Adolescents; Urban; Food Desert; Food Insecurity; Obesity; Baltimore City; Peer mentors; Multi level; Policy; Caregivers; Systems; Agent Based Model; Systems Dynamic Model; Corner Store; Carryout; Recreation Center; Text Messaging; Social Media; Mapping
MeSH Terms: conditions — Obesity | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): The intervention is a multi-level, multi-component intervention designed to increase access to and consumption of healthier foods in low-income, urban, minority neighborhoods. Intervention components will occur at the policy level; food wholesaler level; small food retail outlet level; neighborhood level; household level.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Similar to many community- based public health research programs, the control arm will not receive any intervention components during the initial intervention period. However, after all assessments are completed they will receive a 'delayed intervention' protocol, where the community receives the intervention elements as described in the intervention arm after assessment measures have been completed.

INTERVENTIONS:
Behavioral: Intervention — Intervention components will occur at the policy level (working within Baltimore City policy makers to sustain intervention components, and develop virtual simulations of the Baltimore food environment); food wholesaler level (working with wholesalers to stock healthier food items and provide pricing incentives to storeowners on healthier foods); small food retail outlet level (working with corner store and carry-out owners to stock, promote, and sell healthier foods and beverages); neighborhood level (working with Baltimore college students to deliver nutrition intervention sessions to younger youth in recreation centers in intervention neighborhoods); household level (providing a text messaging and social media program that provides parents and caregivers tips for healthier eating in their respective neighborhoods).
  Arms: Intervention

SUMMARY:
The BHCK study will develop, implement, and evaluate a community-based obesity prevention program, which operates at multiple levels of an urban food system (policy, wholesaler, corner stores, carryout, household, individual; in Baltimore, MD), and will improve the healthy food supply chain to increase affordability, availability, purchasing and consumption of healthy foods within low-income, minority neighborhoods.

DETAILED DESCRIPTION:
Our overarching goal is to develop and evaluate a community-based obesity prevention program, which operates at multiple levels of an urban food system (policy, wholesaler, corner stores, carryout, household, individual; in Baltimore, MD), and will improve the healthy food supply chain to increase affordability, availability, purchasing and consumption of healthy foods within low-income minority neighborhoods. Our research will include stakeholders/ partners at different levels, e.g., the policy, wholesaler, retailer, adult caregiver, and individual child levels, and then develop, implement, and assess a two year multi-level systems-based child obesity prevention strategy targeting minority and low-income children (predominantly AA). Thirty low-income, predominantly AA geographic zones will be identified ("healthy eating zones"). Half of these zones will be randomized to intervention, while the other half will be control. Within each intervention zone we will work with 3-5 small food stores and prepared food sources to increase access to healthy foods through wholesaler discounts, display point of purchase promotional materials, and provide nutrition and food preparation education targeting youth and caregivers. We will work with local policymakers to institutionalize and sustain these changes.

The project will evaluate the impact of the program on: a) healthy food pricing and availability, b) low income African American adult food purchasing and preparation, and c) low-income African American youth diet, and associated psychosocial factors.

ELIGIBILITY:
Inclusion Criteria for Child participants:

9-14 years of age Living within one of the intervention neighborhoods Family does not anticipate moving outside of the study area during the duration of intervention

Inclusion Criteria for Adult Caregiver participants:

Parent/ legal guardian of a child ages 9-14 years of age Living within one of the intervention neighborhoods Family does not anticipate moving outside of the study area during the duration of intervention

Exclusion criteria:

Families that do not have a child within the age range Families that do not live within the neighborhoods in the study area Families who will move outside the study area within the intervention timeframe

Ages: 9 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 890 (Estimated)
Dates: Start 2012-01; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Small Retail Food Store - Healthy Food Availability | Up to 4 years
  A food environment checklist (a modified from the NEMS questionnaire) will be conducted before and after the intervention to assess healthy food availability in both intervention and comparison neighborhoods/ stores.

SECONDARY OUTCOMES:
Household Healthy Food Purchasing | Up to 4 years
  At the adult consumer level, we will use an Adult Impact Questionnaire to examine trends in frequency of purchasing of specific promoted foods pre- and post-intervention. We will score the questionnaire to look at individual food items, as well as at changes in groups of foods developed previously (e.g., healthy and unhealthy food scores, and based on Healthy Eating Index categories).

OTHER OUTCOMES:
Dietary intake of urban, African American youth participants (specifically total calories and fat consumption.) | Up to 4 years
  We will use the Block 2004 Kids Food Frequency questionnaire to assess differences in dietary intake from pre- to post intervention. Data from the FFQ will include total caloric intake and fat intake, along wit other dietary markers.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Gittelsohn, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Coakley HL, Steeves EA, Jones-Smith JC, Hopkins L, Braunstein N, Mui Y, Gittelsohn J. Combining Ground-Truthing and Technology to Improve Accuracy in Establishing Children's Food Purchasing Behaviors. J Hunger Environ Nutr. 2014;9(3):418-430. doi: 10.1080/19320248.2014.898173. PMID 25729465
- [Background] Gittelsohn J, Anderson Steeves E, Mui Y, Kharmats AY, Hopkins LC, Dennis D. B'More Healthy Communities for Kids: design of a multi-level intervention for obesity prevention for low-income African American children. BMC Public Health. 2014 Sep 11;14:942. doi: 10.1186/1471-2458-14-942. PMID 25209072
- [Background] Anderson Steeves E, Martins PA, Gittelsohn J. Changing the Food Environment for Obesity Prevention: Key Gaps and Future Directions. Curr Obes Rep. 2014 Dec;3(4):451-8. doi: 10.1007/s13679-014-0120-0. PMID 25574452
- [Background] Gudzune KA, Welsh C, Lane E, Chissell Z, Anderson Steeves E, Gittelsohn J. Increasing access to fresh produce by pairing urban farms with corner stores: a case study in a low-income urban setting. Public Health Nutr. 2015 Oct;18(15):2770-4. doi: 10.1017/S1368980015000051. Epub 2015 Feb 4. PMID 25649045
- [Background] Gittelsohn J, Mui Y, Adam A, Lin S, Kharmats A, Igusa T, Lee BY. Incorporating Systems Science Principles into the Development of Obesity Prevention Interventions: Principles, Benefits, and Challenges. Curr Obes Rep. 2015 Jun;4(2):174-81. doi: 10.1007/s13679-015-0147-x. PMID 26069864
- [Background] Sattler M, Hopkins L, Anderson Steeves E, Cristello A, Mccloskey M, Gittelsohn J, Hurley K. Characteristics of Youth Food Preparation in Low-Income, African American Homes: Associations with Healthy Eating Index Scores. Ecol Food Nutr. 2015;54(4):380-96. doi: 10.1080/03670244.2014.1001982. Epub 2015 Feb 23. PMID 25706350
- [Background] Vedovato GM, Surkan PJ, Jones-Smith J, Steeves EA, Han E, Trude AC, Kharmats AY, Gittelsohn J. Food insecurity, overweight and obesity among low-income African-American families in Baltimore City: associations with food-related perceptions. Public Health Nutr. 2016 Jun;19(8):1405-16. doi: 10.1017/S1368980015002888. Epub 2015 Oct 6. PMID 26441159
- [Background] Anderson Steeves E, Jones-Smith J, Hopkins L, Gittelsohn J. Perceived Social Support From Friends and Parents for Eating Behavior and Diet Quality Among Low-Income, Urban, Minority Youth. J Nutr Educ Behav. 2016 May;48(5):304-310.e1. doi: 10.1016/j.jneb.2015.12.014. Epub 2016 Feb 8. PMID 26865358
- [Background] Gittelsohn J, Trude A. Environmental Interventions for Obesity and Chronic Disease Prevention. J Nutr Sci Vitaminol (Tokyo). 2015;61 Suppl(Suppl):S15-6. doi: 10.3177/jnsv.61.S15. PMID 26598834
- [Background] Mui Y, Lee BY, Adam A, Kharmats AY, Budd N, Nau C, Gittelsohn J. Healthy versus Unhealthy Suppliers in Food Desert Neighborhoods: A Network Analysis of Corner Stores' Food Supplier Networks. Int J Environ Res Public Health. 2015 Nov 30;12(12):15058-74. doi: 10.3390/ijerph121214965. PMID 26633434
- [Background] Wong MS, Nau C, Kharmats AY, Vedovato GM, Cheskin LJ, Gittelsohn J, Lee BY. Using a computational model to quantify the potential impact of changing the placement of healthy beverages in stores as an intervention to "Nudge" adolescent behavior choice. BMC Public Health. 2015 Dec 23;15:1284. doi: 10.1186/s12889-015-2626-0. PMID 26700158
- [Background] Sato PM, Steeves EA, Carnell S, Cheskin LJ, Trude AC, Shipley C, Mejia Ruiz MJ, Gittelsohn J. A youth mentor-led nutritional intervention in urban recreation centers: a promising strategy for childhood obesity prevention in low-income neighborhoods. Health Educ Res. 2016 Apr;31(2):195-206. doi: 10.1093/her/cyw011. Epub 2016 Mar 2. PMID 26936480
- [Background] Ewart-Pierce E, Mejia Ruiz MJ, Gittelsohn J. "Whole-of-Community" Obesity Prevention: A Review of Challenges and Opportunities in Multilevel, Multicomponent Interventions. Curr Obes Rep. 2016 Sep;5(3):361-74. doi: 10.1007/s13679-016-0226-7. PMID 27379620
- [Derived] Trude ACB, Surkan PJ, Cheskin LJ, Gittelsohn J. A multilevel, multicomponent childhood obesity prevention group-randomized controlled trial improves healthier food purchasing and reduces sweet-snack consumption among low-income African-American youth. Nutr J. 2018 Oct 29;17(1):96. doi: 10.1186/s12937-018-0406-2. PMID 30373597
- [Derived] Trude ACB, Kharmats AY, Jones-Smith JC, Gittelsohn J. Exposure to a multi-level multi-component childhood obesity prevention community-randomized controlled trial: patterns, determinants, and implications. Trials. 2018 May 22;19(1):287. doi: 10.1186/s13063-018-2663-y. PMID 29788977
- See also: Healthy Stores Website — http://www.healthystores.org